CLINICAL TRIAL: NCT01432405
Title: Effect of Exenatide Treatment on Hepatic Fat Content and Plasma Adipocytokine Levels in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect Of Exenatide Treatment on Liver Fat Content in Patients With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mandeep Bajaj, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21068
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone and exenatide (Experimental): Exenatide 10 micrograms injected subcutaneously twice daily plus pioglitazone 45 mg daily orally for 12 months.
  Interventions: Drug: Exenatide; Drug: Pioglitazone
- Pioglitazone (Experimental): Pioglitazone 45 mg daily orally for 12 months
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Exenatide — Type 2 diabetic subjects will be randomized to receive exenatide 10 micrograms injected subcutaneously twice daily for 12 months. Prior to randomization, all subjects will receive baseline measurements of fasting plasma glucose, plasma adipocytokines, Free Fatty Acids, insulin, plasma lipids, and HbA1c as well as measurement of liver fat content with magnetic resonance spectroscopy. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, insulin and adipocytokines as well as hepatic fat content determination at the end of the 12 month treatment period.
  Other Names: Byetta
  Arms: Pioglitazone and exenatide
Drug: Pioglitazone — Type 2 diabetic subjects will be randomized to receive pioglitazone 45 mg daily orally for 12 months. Prior to randomization, all subjects will receive baseline measurements of fasting plasma glucose, plasma adipocytokines, Free Fatty Acids, insulin, plasma lipids, and HbA1c as well as measurement of liver fat content with magnetic resonance spectroscopy. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, insulin and adipocytokines as well as hepatic fat content determination at the end of the 12 month treatment period.
  Other Names: Actos

SUMMARY:
The purpose of this study is to examine the effect of exenatide, an anti-diabetes medication, on liver fat and blood levels of proteins that influence liver fat.

DETAILED DESCRIPTION:
Obesity is characterized as generalized expansion of all adipose tissue depots, an increase in tissue lipid content, and dyslipidemia, insulin resistance, and type 2 diabetes. The adipocyte functions not only as a storage depot for fat but as an endocrine organ that releases hormones in response to specific extracellular stimuli or changes in metabolic status. These secreted proteins, carry out a variety of diverse functions, and they have been referred to collectively as adipokines. The adipokines have been postulated to play important roles in the pathogenesis of insulin resistance, hypertension, disorders of coagulation, dyslipidemia, and glucose intolerance, abnormalities associated with insulin resistance syndrome.

These observations are of considerable interest because recent studies have provided evidence that increased hepatic fat content is an important determinant of hepatic insulin resistance in type 2 diabetic patients. Fatty liver is common in type 2 diabetic patients. The mechanisms responsible for the increase in hepatic fat content are unclear. It has been suggested that fatty liver results from accelerated fatty acid mobilization from expanded visceral fat stores and their deposition in the liver as well as decreased hepatic fatty acid oxidation. Weight loss in humans with Non Alcoholic Fatty Liver Disease (NAFLD) is associated with a decrease in hepatic fat content. In addition, thiazolidinediones have been shown to reduce hepatic fat content and improve hepatic insulin sensitivity in patients with type 2 diabetes as well as in non-diabetic patients with NAFLD. The thiazolidinediones initiate their action by binding the peroxisome proliferator activator receptors (PPAR) , which primarily are located on adipocytes. Treatment of insulin-resistant mice as well as type 2 diabetic patients with insulin sensitizing PPAR activators, such as thiazolidinediones, and increases plasma adiponectin levels. Indirect evidence suggests that adiponectin might mediate some of the insulin-sensitizing effects of PPAR agonists.

Exenatide, a Glucagon Like Peptide-1 (GLP-1) receptor agonist approved for treatment of type 2 diabetes, elicited dose-dependent reductions in body weight in association with improved glycemic control in type 2 diabetic patients. In animal models of obesity, exenatide reduces hepatic fat. However, the effect of exenatide treatment in combination with a thiazolidinedione on liver fat content and plasma adipocytokines levels in patients with type 2 diabetes remains to be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must range in age from 30 to 70 years.
2. Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
3. Patients may be of either sex. Female patients must be non-lactating and must either be at least two years post-menopausal, or be using adequate contraceptive precautions or be surgically sterilized.
4. Patients must meet the American Diabetes Association Criteria for diagnosis of type 2 diabetes mellitus.
5. Patients must be on diet therapy alone and/or metformin treatment (stable dose) and have a fasting plasma glucose concentration between 126 and 260 mg/dl.
6. Patients must have Hematocrit greater than 34%.
7. Subjects whose body weight has been stable (±1 Kg) over the three months prior to study will be included.

Exclusion Criteria:

1, Type 1 diabetes.

2. Fasting plasma glucose greater than 260 mg/dl.

3. Patients must not have received a thiazolidinedione for at least 3 months prior to randomization.

4. Patients must not be on insulin treatment or have received insulin for more than one week within the previous year prior to entry. Patients should not be on sulfonylureas, sitagliptin, or exenatide treatment.

5. Patients taking systemic glucocorticoids or other medications known to affect glucose tolerance are excluded.

6. Patients taking medications that affect gastrointestinal motility will be excluded

7. Patients with a history of Congestive Heart failure (CHF), or clinically significant cardiac, liver or kidney disease (creatinine greater than 1.8 mg/dl).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Bajaj, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Samson SL, Sathyanarayana P, Jogi M, Gonzalez EV, Gutierrez A, Krishnamurthy R, Muthupillai R, Chan L, Bajaj M. Exenatide decreases hepatic fibroblast growth factor 21 resistance in non-alcoholic fatty liver disease in a mouse model of obesity and in a randomised controlled trial. Diabetologia. 2011 Dec;54(12):3093-100. doi: 10.1007/s00125-011-2317-z. Epub 2011 Sep 29. PMID 21956711

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone and Exenatide: Exenatide 10 micrograms injected subcutaneously twice daily plus pioglitazone 45 mg daily orally for 12 months.
  Pioglitazone and exenatide: Type 2 diabetic subjects will be randomized to receive either pioglitazone 45 mg daily orally or exenatide 10 micrograms injected subcutaneously twice daily plus pioglitazone 45 mg daily orally for 12 months. Prior to randomization, all subjects will receive baseline measurements of fasting plasma glucose, plasma adipocytokines, Free Fatty Acids, insulin, plasma lipids, and HbA1c as well as measurement of liver fat content with magnetic resonance spectroscopy. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, insulin and adipocytokines as well as hepatic fat content determination at the end of the 12 month treatment period.
- Pioglitazone: Pioglitazone 45 mg daily orally for 12 months
  Pioglitazone: Type 2 diabetic subjects will be randomized to receive either pioglitazone 45 mg daily orally or exenatide 10 micrograms injected subcutaneously twice daily plus pioglitazone 45 mg daily orally for 12 months. Prior to randomization, all subjects will receive baseline measurements of fasting plasma glucose, plasma adipocytokines, Free Fatty Acids, insulin, plasma lipids, and HbA1c as well as measurement of liver fat content with magnetic resonance spectroscopy. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, insulin and adipocytokines as well as hepatic fat content determination at the end of the 12 month treatment period.
Period: Overall Study
Arm/Group | Pioglitazone and Exenatide | Pioglitazone
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone and Exenatide | Pioglitazone | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (3) | 55 (3) | 52 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fat
Description: The effect of exenatide and pioglitazone on liver fat content after one year of treatment in patients with type 2 diabetes.
Time Frame: one year
Measure: Mean (Standard Error); unit: percent of liver fat
Arm/Group | Pioglitazone and Exenatide | Pioglitazone
Number analyzed (Participants) | 11 | 10
percent of liver fat | 4.7 (1.3) | 6.5 (1.9)

2. Secondary Outcome: Plasma Adipocytokines
Description: the effect of the intervention on plasma adiponectin levels.
Time Frame: one year
Measure: Mean (Standard Error); unit: microgram per ml
Arm/Group | Pioglitazone and Exenatide | Pioglitazone
Number analyzed (Participants) | 11 | 10
microgram per ml | 23.2 (2.7) | 15.8 (1.4)

ADVERSE EVENTS:
Arm/Group | Pioglitazone and Exenatide | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes